CLINICAL TRIAL: NCT04299568
Title: Effects of Anti-gravity Treadmill Training on Knee Osteoarthritis in Geriatric Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Collaborators: Higher Education Commission (Pakistan) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/1
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor who will be responsible for collecting the data from the participants in the study will be unaware to the allocation of the participants to the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti gravity treadmill training (Experimental): Heat Therapy in combination with Electro-therapy for 10 minutes, followed by tibio-femoral and patello-femoral joint mobilization followed by Lower Body Positive Pressure (LBPP) treadmill training for 15 minutes.
  Interventions: Device: Anti gravity treadmill training; Procedure: Physical Therapy
- Control (Active Comparator): Heat Therapy in combination with Electro-therapy for 10 minutes, followed by tibio-femoral and patello-femoral joint mobilization only
  Interventions: Procedure: Physical Therapy

INTERVENTIONS:
Device: Anti gravity treadmill training — Lower Body Positive Pressure (LBPP) treadmill training for 15 minutes
  Other Names: Lower Body Positive Pressure (LBPP) treadmill training
  Arms: Anti gravity treadmill training
Procedure: Physical Therapy — Heat Therapy in combination with Electro-therapy for 10 minutes, followed by tibio-femoral and patello-femoral joint mobilization

SUMMARY:
Knee osteoarthritis is a very common disorder affecting majority of elderly population. There is considerable functional disability associated with this disorder. The financial burden associated with this disease is quite high. Although various forms of pharmacologic and non pharmacologic therapies exist for its management, but most of these interventions only deal with symptoms without taking into account the associated factors aggravating the condition. Research suggests that abnormal loading of an arthritic joint will only increase the pain and disability. Participation in a regular exercise program involving weight bearing activities is a successful way to reduce or prevent decline in functional abilities. But the major problem with this approach lies in its abnormal loading of joint leading to altered biomechanics resulting in more joint damage. To counter this problem, lower body positive pressure or anti gravity treadmills have been designed. These treadmills provide up to 80% body weight support, thus considerably un-weighing the joint while retaining proper joint biomechanics. So with the help of this specialized training unit, elderly population will be better equipped to cope with arthritic changes leading to greater functional independence.

DETAILED DESCRIPTION:
Osteoarthritis is a very common chronic joint disease resulting in functional disability. Knee OA is considered to be most common form of arthritis in western countries. Knee OA is mainly characterized by presence of pain, radiographic evidence of reduced joint space, wear and tear of articular cartilage and formation of osteophytes i.e., new bone formation at the center and margins of joint. Pain and resultant joint changes causes a change in joint biomechanics and an eventual disuse of limb leading to muscle weakness and atrophy. According to an estimate from a study, knee OA nearly affects 10% of people older than 55 years of age, resulting in severe functional disability in a quarter of this affected population. In elderly population, knee OA poses almost the same risk of disability as caused by heart disease and a larger threat than due to any other medical condition. The prevalence of OA is reported to be as high as 28% in urban and 25% in rural areas of Pakistan.

Literature on knee OA treatment suggest that weight bearing activities in the form of walking are useful in the management of joint symptoms. Loading across the joint must be optimal so that there is no abnormal stress on any compartment of the joint. Abnormal valgus and varus stress results in 4 fold and 5 fold increase in lateral and medial compartments OA of the knee respectively. But this increased loading on an already worn joint can cause considerable pain and damage to the joint. For this purpose, aquatic exercises and hydrotherapy are usually used to counteract the forces acting on the joint. Then there are different types of harness systems and robotic devices to physically lift the patients for unloading the joint. But the problem with these interventions is that they do not account for proper joint kinematics necessary for optimal distribution of forces across the joints. For this purpose, anti gravity treadmills or lower body positive pressure treadmills are designed which take into account the proper joint kinematic s while partially un-weighing the joint. These treadmills are based on NASA technology used for astronauts to counteract the joint problems experienced by them.

These treadmills consist of an air tight chamber surrounding the lower body in which increased pressure is applied, so that the treadmill causes an upward lifting force. This results in successfully decreasing the body weight and gravitational forces on the lower extremity to an adjustable level with a high degree of consistency. Body weight can then be adjusted to as small increments as 1% and as large as 80% by using positive air pressure. This method is considered superior to other methods of un-weighing (harness systems and aquatic therapy) because there is uniform application of pressure over the lower limbs, thereby decreasing the creation of pressure points (common with harness systems) while retaining normal muscle activation and gait patterns (which are changed during water based activities).

This study will help the patients suffering from osteoarthritis to rehabilitate in a pain free environment focusing on proper joint kinematics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age group 50-75 years
* Knee osteoarthritis GI, GII and G III (Kellgren & Lawrence system).

Exclusion Criteria:

* Traumatic arthritis
* Unstable cardiovascular state
* Neuro-muscular disorders involving the lower extremity
* History of surgery of lower limb

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  Numeric Pain Rating Scale will be used to measure patient's self perceived pain.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | 4 weeks
  Knee Injury and Osteoarthritis Outcome Score will be used to assess patients symptoms, physical functioning and quality of life.
36-Item Short Form Survey for Quality of Life | 4 weeks
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures

CONTACTS AND LOCATIONS:
Overall Officials: Aamer Naeem, BSPT, PPDPT, MSOMPT, PhD*, Principal Investigator — Foundation University Islamabad; Muhammad Osama, DPT, MSOMPT, CHPE, ACMEd, PhD*, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Heer HD, Kaufman A, Repka CP, Rojas K, Charley B, Bounds R. AlterG Anti-Gravity Treadmill Accuracy of Unloading Is Affected by Support Frame Height. J Strength Cond Res. 2021 Oct 1;35(10):2910-2914. doi: 10.1519/JSC.0000000000003223. PMID 31403571
- [Background] Liang J, Guo Y, Zheng Y, Lang S, Chen H, You Y, O'Young B, Ou H, Lin Q. The Lower Body Positive Pressure Treadmill for Knee Osteoarthritis Rehabilitation. J Vis Exp. 2019 Jul 22;(149). doi: 10.3791/59829. PMID 31380828
- [Background] Liang J, Lang S, Zheng Y, Wang Y, Chen H, Yang J, Luo Z, Lin Q, Ou H. The effect of anti-gravity treadmill training for knee osteoarthritis rehabilitation on joint pain, gait, and EMG: Case report. Medicine (Baltimore). 2019 May;98(18):e15386. doi: 10.1097/MD.0000000000015386. PMID 31045790
- [Background] Peeler J, Leiter J, MacDonald P. Effect of Body Weight-Supported Exercise on Symptoms of Knee Osteoarthritis: A Follow-up Investigation. Clin J Sport Med. 2020 Nov;30(6):e178-e185. doi: 10.1097/JSM.0000000000000668. PMID 30277892
- [Background] Peeler J, Ripat J. The effect of low-load exercise on joint pain, function, and activities of daily living in patients with knee osteoarthritis. Knee. 2018 Jan;25(1):135-145. doi: 10.1016/j.knee.2017.12.003. Epub 2018 Jan 8. PMID 29325839
- [Background] Bugbee WD, Pulido PA, Goldberg T, D'Lima DD. Use of an Anti-Gravity Treadmill for Early Postoperative Rehabilitation After Total Knee Replacement: A Pilot Study to Determine Safety and Feasibility. Am J Orthop (Belle Mead NJ). 2016 May-Jun;45(4):E167-73. PMID 27327921
- [Background] Peeler J, Christian M, Cooper J, Leiter J, MacDonald P. Managing Knee Osteoarthritis: The Effects of Body Weight Supported Physical Activity on Joint Pain, Function, and Thigh Muscle Strength. Clin J Sport Med. 2015 Nov;25(6):518-23. doi: 10.1097/JSM.0000000000000173. PMID 25647537